CLINICAL TRIAL: NCT06551454
Title: Smart Textile Solutions as Biofeedback Method for Injury Prevention for Latvian Football Youth League Players
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riga Stradins University (Other)
Responsible Party: Principal Investigator, Guna Semjonova, Dr. Principal Investigator, Scientific Project Coordinator, Department of Rehabilitation at Riga Stradins University, Riga Stradins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: lzp-2023/1-0027
Record Dates: First submitted 2024-07-24; First posted 2024-08-13 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Sport Injury
Keywords: smart textile sock system; youth athletes; football; soccer; biofeedback; injurie prevention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Football Youth League Players group (Active Comparator): Intervention for all participants: 12 weeks of prevention exercise program in football FIFA 11+ tasks of part 2: single leg stance and squats. Followed by exercise monitoring instructions in the FIFA 11+ user manual.
  Interventions: Device: Smart Textile Solution Biofeedback Method
- Smart Textile Biofeedback Football Youth League Players group (Experimental): Using the biofeedback method provided by the DAid® smart sock system as the monitoring method of positioning the lower limb for the study group during 12 weeks of prevention exercise program in football FIFA 11+ tasks of part 2: single leg stance and squats.
  Interventions: Device: Smart Textile Solution Biofeedback Method

INTERVENTIONS:
Device: Smart Textile Solution Biofeedback Method — The Smart Textile Solution Biofeedback Method for injury prevention in youth league football players integrates sensors within socks to monitor key biomechanical indicators such as center of pressure and plantar pressure of the foot in real-time. By providing immediate feedback and alerts on potential injury risks, the system helps players adjust their techniques during training sessions and prevent injuries during training and games.

SUMMARY:
Lower limb injuries are the most common in youth football leagues, accounting for 72% to 93% of all injuries. The leading prevention program in football today is the FIFA 11+ warm-up program, which reduces the risk of injury by 30%. Evidence from several studies confirms the addition of feedback during training reduces the incidence of injury by 40% . Recent studies have shown that the smart textile sock system is an objective, easy-to-use tool for real-time foot monitoring and is an interactive feedback tool for athletes. However, there is a lack of information on the impact of the objective feedback provided by the Smart Textile Sensor Socks System on the outcome measures of football players prevention programs. In the first phase of the project, a cross-sectional study involving youth league footballers will be conducted to identify the most effective feedback elements of the smart sock system. In the second phase, a pilot study will be conducted to evaluate the effectiveness of prevention exercises using the feedback provided by smart textile sensor socks. The results of the functional tests and the study outcomes will be selected as performance indicators to evaluate the smart textile sensor sock system. Conclusions on the use of the smart textile sensor sock system as a feedback method for injury prevention in Latvian Youth Football League players will be drawn based on the results obtained from the project.

ELIGIBILITY:
Inclusion Criteria:

1. youth football league players;
2. agree to participate in the study;
3. age from 14 to 18 years;
4. understands and speaks Latvian.

Exclusion Criteria:

1. operative treatment in the lower limb within the last 9 months;
2. injuries or pain in the lower limb during the last 6 months;
3. disorders of the vestibular apparatus
4. presence of metallic implants in the sensor application areas.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Foot plantar pressure changes during functional tasks (FIFA 11+; Part 2) | 12 weeks
  Data from the biofeedback method provided by the biofeedback DAid® smart sock system
Functional Movement | 2 times: pre and post 12 week intervention
  Change of Functional Movement Screening (FMS™) Scores

SECONDARY OUTCOMES:
Age | 1 time.
  Age in years
Sex | 1 time
  Answers: male, female
Foot size | 1 time
  By using In the Continental European system, where the shoe size is the length of the last, expressed in Paris points or 2⁄3 cm (6.67 mm), for both sexes and for adults and children alike. The Continental European system is used in Austria, Belgium, Denmark, France, Germany, Italy, Luxembourg, the Netherlands, Norway, Poland, Portugal, Spain, Sweden, Switzerland and most other continental European countries such as Latvia. The system is sometimes described as Stich size (from Pariser Stich, the German name for the Paris point), or Stichmaß size (from a German name of a micrometer for internal measurements). Shoe/ Stichmaß size 32 - 48.
positions on football field | 1 time
  1 - Goalkeeper · 2 - Right Back · 3 - Left Back · 4 - Center Back · 5 - Center Back · 6 - Defensive Midfield · 7 - Right Wing/Forward · 8 - Central Midfield.
User experience | Once - after 12 weeks of intervention
  Evaluated by System Usability Scale scale, user motivation intrinsic scale. The system usability scale (SUS) is a simple, ten-item attitude Likert scale giving a global view of subjective assessments of usability. The usability of a system, as defined by the ISO standard ISO 9241 Part 11, can be measured by taking into account the context of use of the system-i.e., who is using the system, what they are using it for, and the environment in which they are using it. Furthermore, measurements of usability have several different aspects: - effectiveness (can users successfully achieve their objectives); - efficiency (how much effort and resource is expended in achieving those objectives); - satisfaction (was the experience satisfactory). The formula for computing the final SUS score requires converting the raw scores, by subtracting 1 from each raw score, then utilizing the equation.
Frequency of non-contact injuries (predicted number of injuries) | 1 year after 12-weeks intervention
  A one-year follow-up of records of the Frequency of non-contact injuries (predicted number of injuries)

CONTACTS AND LOCATIONS:
Overall Officials: Signe Tomsone, Dr.Med., Principal Investigator — Faculty of Health and Sports Sciences, Department of Rehabilitation, Riga Stradiņš University; Linda Lancere, Dr.sc.ing., Principal Investigator — Vidzeme University of Applied Sciences; Aleksejs Katasevs, Dr.phys, Principal Investigator — Riga Technical University; Aleksandrs Okss, Dr.Habil.Sci-Eng., Principal Investigator — Riga Technical University
Locations (1):
- Latvian Football Federation, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No
https://zenodo.org/records/12804841

REFERENCES:
- See also: Following link is for the data management plan description of the project titled "Smart Textile Solutions as Biofeedback Method for Injury Prevention for Latvian Football Youth League Players" — https://zenodo.org/records/12804841